CLINICAL TRIAL: NCT01766726
Title: Effects of Newly-Initiated QUAD Therapy on Aortic/Coronary Inflammation in ART-Naïve Infected Patients
Acronym: Quad
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2012P001138
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: HIV
Keywords: HIV; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy control subjects: Historical healthy control subjects matched to HIV+ patients on traditional cardiovascular risk factors will be studied at baseline with respect to arterial inflammation and coronary atherosclerotic plaque. Prospectively recruited healthy control subjects matched to HIV+ patients on traditional cardiovascular risk factors will be studied at baseline with respect to lipid and immune function.
- ART-naïve HIV+ patients starting QUAD/Stribild: ART-naïve HIV+ patients who are about to be started QUAD/Stribild by their treating clinicians will be studied at baseline and 6 months after initiating QUAD/Stribild therapy.

SUMMARY:
The main aims of this study are to determine whether: a) ART-naïve HIV+ subjects have increased artherosclerotic plaque inflammation/vulnerability, b) newly-initiated QUAD/Stribild therapy will decrease plaque inflammation/vulnerability in these subjects, and c) QUAD/Stribild therapy will improve indices of immune dysregulation and lipid dysfunction as a mechanism of improved plaque inflammation/vulnerability. Parameters of lipid and immune function will also be assessed in healthy control subjects, for comparison.

DETAILED DESCRIPTION:
Patients with HIV are at higher risk of morbidity and mortality from cardiovascular disease than healthy subjects. Antiretroviral therapy (ART) has greatly increased the lifespan of HIV+ patients, but their risk of CVD remains higher than normal. Previously, it has been shown that compared to healthy control subjects, ART-treated HIV+ patients have more atherosclerotic plaque inflammation in the aorta. This study is intended to determine whether atherosclerotic plaque inflammation/vulnerability is increased in ART-naïve HIV+ patients and whether these parameters can be improved through 6 months of newly-initiated QUAD/Stribild therapy. Additionally, the study will determine whether indices of immune dysregulation and lipid dysfunction are increased in ART-naive HIV+ patients and whether these parameters can also be improved through 6 months of newly initiated QUAD/Stribild therapy.

ELIGIBILITY:
HIV-infected Subjects:

Inclusion Criteria:

* men and women, ages 18+, with documented HIV-infection who are ART-naive and ready to be started on ART with QUAD/Stribild by their treating infectious disease doctors

Exclusion Criteria:

* history of prior, sustained ART use
* CD4 <50 or AIDS-defining illness
* known current opportunistic infection or acute infections (not including Hepatitis B/C)
* pregnancy or breastfeeding
* history of acute coronary syndrome or coronary artery stenting or surgery, diabetes mellitus, or significant autoimmune/inflammatory disease
* plans for sustained use during 6 month study interval of a confounding immune suppressant medication including intravenous or oral corticosteroid
* hemoglobin < 12.5 g/dl for men or < 12 g/dl for women
* eGFR < 70 ml/min/1.73 m2 calculated by CDK-EPI
* contrast dye allergy
* contraindication to beta blockers or nitroglycerin administered during MDCT coronary angiography (coronary CTA) protocol
* body weight > 320 lbs (PET scanner limitation)
* significant radiation exposure (>2 myocardial perfusion scans or CT angiograms) received within the past year
* reported active illicit drug use

Healthy control subjects:

Inclusion Criteria:

-men and women, ages 18+, without HIV infection

Exclusion Criteria:

* known current opportunistic infection or acute infections (not including Hepatitis B/C)
* pregnancy or breastfeeding
* history of acute coronary syndrome or coronary artery stenting or surgery, diabetes mellitus, or significant autoimmune/inflammatory disease
* sustained use of a confounding immune suppressant medication including intravenous or oral corticosteroid
* hemoglobin < 12.5 g/dl for men or < 12 g/dl for women
* reported active illicit drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with HIV infection being cared for in the Eastern Massachusetts area may be appprised of the study by their treating infectious disease doctors. Additionally, subjects with HIV infection from the community will be recruited via posters, advertisements, e-postings. Healthy control subjects from the community will be recruited via posters, advertisements, and e-postings.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Aortic/coronary target to background ratio (TBR) on cardiac FDG-PET | Baseline and change from baseline to 6 months in HIV cohort starting QUAD/Stribild
  Degree of aortic/coronary atherosclerotic plaque inflammation assessed via cardiac FDG-PET as target to background ratio (TBR) of the standardized uptake value (SUV).

SECONDARY OUTCOMES:
Aortic/coronary atherosclerotic plaque on coronary computed tomography angiography (coronary CTA) | Baseline and change from baseline to 6 months in HIV cohort starting QUAD/Stribild
  Aortic/coronary atherosclerotic plaque assessed via coronary CTA.
Lipid and lipoprotein levels | Baseline and change from baseline to 6 months in HIV cohort starting QUAD/Stribild
  Levels of lipids and lipoproteins including but not limited to levels of total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, and levels select apolipoprotein levels.
Indices of pro-atherogenic lipid dysfunction | Baseline and change from baseline to 6 months in HIV cohort starting QUAD/Stribild
  Including HDL oxidative potential and other assessments of HDL function and structure.
Inflammatory biomarker levels | Baseline and change from baseline to 6 months in HIV cohort starting QUAD/Stribild
  Levels of inflammatory biomarkers including but not limited to soluble CD163.
Percentage of circulating activated leukocyte subsets | Baseline and change from baseline to 6 months in HIV cohort starting QUAD/Stribild
  Percentage of circulating activated leukocyte subsets including but not limited to percentage of circulating CD14+CD16+ monocytes assessed via flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Toribio M, Burdo TH, Fulda ES, Cetlin M, Chu SM, Feldpausch MN, Robbins GK, Neilan TG, Melbourne K, Grinspoon SK, Zanni MV. Effects of Integrase Inhibitor-Based ART on the NLRP3 Inflammasome Among ART-Naive People With HIV. Open Forum Infect Dis. 2020 Sep 29;7(10):ofaa459. doi: 10.1093/ofid/ofaa459. eCollection 2020 Oct. PMID 33134423
- [Derived] Toribio M, Park MH, Zanni MV, Robbins GK, Burdo TH, Williams KC, Feldpausch MN, Stone L, Melbourne K, Grinspoon SK, Fitzgerald ML. HDL Cholesterol Efflux Capacity in Newly Diagnosed HIV and Effects of Antiretroviral Therapy. J Clin Endocrinol Metab. 2017 Nov 1;102(11):4250-4259. doi: 10.1210/jc.2017-01334. PMID 28945911